CLINICAL TRIAL: NCT03385512
Title: Improving Patient-Centered Communication in Primary Care: A Cluster Randomized Controlled Trial of the Comparative Effectiveness of Three Interventions
Brief Title: OPEN & ASK: Improving Patient-Centered Communication in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Reliant Medical Group (Other); University of Massachusetts, Worcester (Other); Palo Alto Medical Foundation (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Ming Tai-Seale, PhD, MPH, Professor of Family Medicine and Public Health, and Director of Outcomes Analytics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IHS-1608-35689
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Patient Engagement; Physician's Role; Physician-Patient Relations; Patient Activation
Keywords: Virtual standardized patient coaching; Standardized patient instructor coaching; Patient centered communication
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Patient and health care team participants and the clinics in which they practice will be randomly assigned to one of three groups for the duration of their participation in the study: 1) OPEN High Tech, 2) OPEN High Touch and 3) ASK. Unit of randomization is clinic. Physicians will be clustered in clinics and patients clustered within physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OPEN High Touch (Experimental): Participants in this arm will experience the OPEN High Touch intervention.
  Interventions: Behavioral: OPEN High Touch
- OPEN High Tech (Experimental): Participants in this arm will experience the OPEN High Tech intervention.
  Interventions: Behavioral: OPEN High Tech
- ASK Poster (Experimental): Participants in this arm will experience the ASK intervention.
  Interventions: Behavioral: ASK Poster in Exam Rooms

INTERVENTIONS:
Behavioral: OPEN High Touch — This arm will contain three components: (a) a pre-visit questionnaire delivered through the patient portal of the EHR, asking patients what they most want to discuss with their physician in the upcoming visit; (b) an animated video for patients providing coaching on how to best prepare for their upcoming visits and get the most from the visits; and (c) Standardized Patient Instructor (SPI) providing communication coaching for physicians on how to incorporate what matter most to patients in the visit, with empathy, and clarity.
  Arms: OPEN High Touch
Behavioral: OPEN High Tech — The patient components of the intervention will be identical to the patient components of the High Touch arm (i.e., the pre-visit survey and patient coaching video). The difference will be in the PCP training: we will replace the in-person SPI with a mobile app program.
  Arms: OPEN High Tech
Behavioral: ASK Poster in Exam Rooms — This arm is intended to activate patients by encouraging them to ask three questions during their primary care visit: (1) What are my options? (2) What are the possible benefits and risks of each option? (3) How likely are the benefits and risks of each option to occur to me? This will involve placing posters with these questions in all exam rooms used by providers in clinics randomized to the ASK arm of the trial.
  Arms: ASK Poster

SUMMARY:
This large scale multi-center cluster randomized controlled trial (RCT) is designed to assess the comparative effectiveness of three interventions in diverse ambulatory care settings and patient populations. Findings will help healthcare systems decide which approach to adopt to empower patients and enable providers to engage in patient centered communication. The specific aims are to:

1. Engage with patients and healthcare providers who have used the tools in the pilot study (ClinicalTrials.gov Identifier NCT02522286) at the Sutter Health Palo Alto Medical Foundation (PAMF), as well as new stakeholders at University of California San Diego Health System and Meyers Primary Care Institute at University of Massachusetts and Reliant Medical Group, to further refine and adapt these patient-centered interventions to be integrated into real world primary care clinics.
2. Conduct a large scale cluster RCT with three arms, to evaluate the comparative effectiveness of three interventions: OPEN with in-person SPI training (High Touch), OPEN with online SPI training (High Tech), and ASK. Primary outcomes will include patient perceptions of how well their PCPs have engaged them in patient centered communication. The investigators will also measure patients' confidence in managing their health, intention to follow through with care plans, and downstream behaviors in following through with care plans, use of services such as phone calls, secure messaging, and additional visits.
3. Identify the strategy that has the most potential for sustained impact and replication within and across healthcare systems. The investigators will analyze the fidelity to the intervention protocols, including consistency of delivery as intended and the time/effort involved in implementing the interventions. The investigators will also assess the extent to which the programs become institutionalized.

The investigators anticipate that this multi-level healthcare system intervention will result in significant improvement in: patient satisfaction with how PCP has engaged them in the visit, confidence in selfcare; patients' intention to adhere to care plan, and clinical indicators. Furthermore, more effective communication would lower health service utilization after the visit. The investigators further expect that the intervention will affect physicians', medical assistants' and nurses' experience as well as healthcare system leaders' intention to implement in routine practice.

DETAILED DESCRIPTION:
This is a three-arm, multi-site, cluster-randomized controlled trial, comparing three approaches to improve communication between patients and their doctors. Three health systems will participate in the study: UCSD Health, Reliant Medical Group, and Sutter Health.

The study will be carried out in 2 phases.

Phase 1: Phase 1 includes intervention and survey development work to take place prior to the RCT.

OPEN High Touch intervention - The High Touch intervention will be modeled after the Open Communication intervention developed in the pilot (ClinicalTrials.gov Identifier NCT02522286) which contained three components: (a) a one question pre-visit survey delivered through the patient portal of the EHR, asking patients what they most want to discuss with their physician in the upcoming visit; (b) an animated video for patients providing coaching on how to best prepare for their upcoming visits and get the most from the visits; and (c) Standardized Patient Instructor (SPI) providing communication coaching for physicians on how to incorporate what matter most to patients in the visit, with empathy, and clarity.

OPEN High Tech intervention - For the High Tech arm, the patient components of the intervention will be identical to the patient components of the High Touch arm (i.e., the pre-visit survey and patient coaching video). The difference will be in the PCP training: we will replace the in-person SPI with a mobile app with embedded audio and video vignettes demonstrating the communication challenges (e.g., patient with a big list of issues, patients who resist physician recommendations, and patients who disagree with physician) and recommended strategies. A mobile app offers several advantages, including being accessible at a convenient time for busy providers, being easily disseminated, and easily updated. The app will be interactive, posing questions to learners in association with video vignettes and asking learners to answer how they would handle the situation. We will start with the idea of building a set of short mobile modules that mirror the High Touch approach, honing skills on acknowledging patient's agenda, negotiate a joint agenda, invite patient to teachback and incorporate it in the After Visit Summary in the EHR.

ASK intervention - The ASK intervention is intended to activate patients by encouraging them to ask three questions during their primary care visit: (1) What are my options? (2) What are the possible benefits and risks of each option? (3) How likely are each of the benefits and risks to happen to me? These questions will be printed on posters and placed in exam rooms used by providers in clinics randomized to the ASK arm of the trial.

Phase 2: Phase 2 covers the trial recruitment, and three waves of data collection. Prior to the start of the RCT we will collect baseline (T0) data to allow measurement of primary care provider (PCP) performance prior to the trial. Patients participating in the T0 phase will provide only post-visit ratings of their encounters; we will not collect other outcome data or clinical indicators for these patients. For all patients in the intervention phase, we will be collecting information at two time points: 1) immediately post-encounter (T1); and 2) three months post-encounter (T2). We will further sample the top 5% high users of services after the intervention and review their medical records including the indexed visit and subsequent services that had occurred within four weeks after the indexed visit. The chart review will enable us to decipher the reasons for high volume of services after the indexed visit. We will also use existing patient survey data (Press-Ganey and/or NRC) to supplement our data sources.

Analytical approach: We will apply intention to treat analysis, providing descriptive statistics on relevant outcome measures across patients, PCPs, and clinics according to their randomized assignments in the RCT. We will then use generalized estimating equations logistic regression analysis to examine the impact of the assignment into the intervention arms and the outcomes, while controlling for patient and physician covariates.

ELIGIBILITY:
Inclusion Criteria:

For patient participants:

* Adults 18 years and older,
* Have an activated account to the patient portal of the electronic health record
* Able to read/write in English or Spanish
* Have an appointment with their PCP, who has volunteered to be participate in the study, during the data collection period
* Willing and able to provide informed consent and complete brief questionnaires online.

For health care team (primary care providers, nurse and medical assistants) participants:

* Employed at one of the participating study clinics
* Willing and able to provide informed consent and complete brief questionnaires online.

Exclusion Criteria:

For patient participants:

* People who don't speak English or Spanish
* People who do not have an active My Chart/My Health Online account.
* Younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5565 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Patient reported experience with care: CollaboRATE | Within 7 days of a regularly scheduled appointment (the indexed visit) and 3 months after the indexed visit.
  Responses from CollaboRATE, a validated 3-item, patient-reported measure of shared decision making compared between baseline and intervention patients; immediately after the indexed visit and 3 months after the indexed visit with their PCP for intervention patients; and across interventions for variations. The 3 questions, which will be answered on a scale of o "No effort was made" to 9 "Every effort was made" are:
  1. How much effort was made to help you understand your health issue?
  2. How much effort was made to listen to the things that matter most to you about your health issues? 3. How much effort was made to include what matters most to you in choosing what to do next?
Patient reported experience with care: Doctor Facilitation subscale of the Perceived Involvement in Care Scale | Within 7 days of a regularly scheduled appointment (the indexed visit) and 3 months after the indexed visit.
  Responses from this validated 5-item, patient reported measure of their perceptions of how well their physician facilitated their involvement in decision making are compared between baseline and intervention patients; immediately after the indexed visit with their PCP and 3 months after the indexed visit for intervention patients; and across interventions for variations. The 5 questions, which will answered on a scale of 0 "Definitely Disagree" to 9 "Definitely Agree" are:
  1. My doctor asked me whether I agree with his/her decisions
  2. My doctor gave me a complete explanation for my medical symptoms or treatment
  3. My doctor asked me what I believe is causing my medical symptoms
  4. My doctor encouraged me to talk about personal concerns related to my medical symptoms
  5. My doctor encouraged me to give my opinion about my medical treatment.

SECONDARY OUTCOMES:
Action Plan | This will be measured within 7 days of the indexed appointment for intervention patients.
  The "Patient Instructions" field of the After Visit Summary that patients receive in paper and/or through their online patient portal after the indexed visit with their provider.
Patient reported confidence to adhere to action plan | This will be measured within 7 days and again 3 months after the indexed visits for intervention patients.
  Responses from a patient reported measure of their confidence to adhere to their action plan. This will be measured by the question "Overall, how confident are you about your ability to take good care of your health?" using a 5-point Likert scale from 1=not confident at all to 5=Completely confident. This is a question used in the Health Information National Trends Survey (HINTS), a biennial, cross-sectional survey of a nationally-representative sample of American adults, developed and used by the Center for Disease Control and Prevention and National Cancer Institute (https://www.healthypeople.gov/2020/data-source/health-information-national-trends-survey).
Patient reported intention to adhere to action plan | This will be measured within 7 days and again 3 months after the indexed visits for intervention patients.
  Responses from this patient reported measure of intention to adhere to their action plan. We will examine the psychometric property of these measures and expect that they will enable us to form a factor that measures the construct of intention to adhere to care plans. We call this measure INTENTION.
Adherence to action plans | This will be measured within 7 days and again 3 months after the indexed visits for intervention patients.
  A patient reported measure that will be adapted from the Medical Outcomes Study (MOS) general adherence survey instrument with help from our study stakeholders.
The Veterans RAND 12-item health survey (VR12) | This will be measured within 7 days and again 3 months after the indexed visits for intervention patients.
  A 12-item patient reported health status measure.
Blood pressure | 12 months after indexed visits for intervention patients.
  This will be extracted from the electronic health record and used as a clinical indicator of health outcomes.
A1c | 12 months after indexed visits for intervention patients.
  This will be extracted from the electronic health record and used as a clinical indicator of health outcomes.
LDL | 12 months after indexed visits for intervention patients.
  This will be extracted from the electronic health record and used as a clinical indicator of health outcomes.
Patient-initiated calls | 12 months after indexed visits for intervention patients.
  These will be measured using structured fields in the electronic health record and access log. The investigators will review the charts of the top 5% of telephone callers.
E-messages | 12 months after indexed visits for intervention patients.
  These will be measured using structured fields in the electronic health record and access log. The investigators will review the charts of the top 5% of e-message senders.
Office visits | 12 months after indexed visits for intervention patients.
  These will be measured using structured fields in the electronic health record. The investigators will review the charts of the top 5% of office visit generators.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Tai-Seale, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - Palo Alto Medical Foundation Research Institute, Mountain View, California
  - University of California San Diego Health System, San Diego, California
  - Meyers Primary Care Institute at University of Massachusetts Medical School/Reliant Medical Group, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
We will make a complete, cleaned, de-identified copy of the final data set used in conducting the final analyses available within 9 months after the completion of the study. Researchers interested in replicating our methods and study findings will have full access to the study protocol, samples of intervention prototypes, analytic methods and codebook. We will deliver our final protocol, prototypes, toolkit, codebook documents, and instructions regarding how other researchers can access our study documents to PCORI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 9 months after the completion of the study.
Access Criteria: A Data Use Agreement will be implemented for other researchers interested in using our data for replication of research findings or for additional areas of research. We will request that outside investigators discuss their manuscript ideas with the PI (Dr. Tai-Seale) and Site-PIs (Dr. Cheryl Stults and Dr. Kathy Mazor) before proceeding. Furthermore, we will request that manuscripts using data from our project be approved by the PI and Site-PIs prior to submission for publication. Members of this project team may contribute as co-authors when data from this study are used. We will request that manuscripts, abstracts, presentations, and chapters developed by other investigators credit this study and credit PCORI as the funding source for the data. This process will allow for a central repository and access point for all papers, abstracts, posters, and presentations by any individual or organization using our data.

REFERENCES:
- [Background] Tai-Seale M, Elwyn G, Wilson CJ, Stults C, Dillon EC, Li M, Chuang J, Meehan A, Frosch DL. Enhancing Shared Decision Making Through Carefully Designed Interventions That Target Patient And Provider Behavior. Health Aff (Millwood). 2016 Apr;35(4):605-12. doi: 10.1377/hlthaff.2015.1398. PMID 27044959
- [Background] Tai-Seale M, Sullivan G, Cheney A, Thomas K, Frosch D. The Language of Engagement: "Aha!" Moments from Engaging Patients and Community Partners in Two Pilot Projects of the Patient-Centered Outcomes Research Institute. Perm J. 2016 Spring;20(2):89-92. doi: 10.7812/TPP/15-123. Epub 2016 Feb 22. PMID 26909777
- [Background] Dillon EC, Stults CD, Wilson C, Chuang J, Meehan A, Li M, Elwyn G, Frosch DL, Yu E, Tai-Seale M. An evaluation of two interventions to enhance patient-physician communication using the observer OPTION5 measure of shared decision making. Patient Educ Couns. 2017 Oct;100(10):1910-1917. doi: 10.1016/j.pec.2017.04.020. Epub 2017 May 1. PMID 28532861
- [Derived] Tai-Seale M, Cheung M, Vaida F, Ruo B, Walker A, Rosen RL, Hogarth M, Fisher KA, Singh S, Yood RA, Garber L, Saphirak C, Li M, Chan AS, Yu EE, Kallenberg G, Longhurst CA, Millen M, Stults CD, Mazor KM. Patient-Clinician Communication Interventions Across Multiple Primary Care Sites: A Cluster Randomized Clinical Trial. JAMA Health Forum. 2024 Dec 6;5(12):e244436. doi: 10.1001/jamahealthforum.2024.4436. PMID 39671203
- [Derived] Stults CD, Mazor KM, Cheung M, Ruo B, Li M, Walker A, Saphirak C, Vaida F, Singh S, Fisher KA, Rosen R, Yood R, Garber L, Longhurst C, Kallenberg G, Yu E, Chan A, Millen M, Tai-Seale M. Patients' Perspectives on Plans Generated During Primary Care Visits and Self-Reported Adherence at 3 Months: Data From a Randomized Trial. J Particip Med. 2024 Mar 14;16:e50242. doi: 10.2196/50242. PMID 38483458
- [Derived] Tai-Seale M, Rosen R, Ruo B, Hogarth M, Longhurst CA, Lander L, Walker AL, Stults CD, Chan A, Mazor K, Garber L, Millen M. Implementation of Patient Engagement Tools in Electronic Health Records to Enhance Patient-Centered Communication: Protocol for Feasibility Evaluation and Preliminary Results. JMIR Res Protoc. 2021 Aug 26;10(8):e30431. doi: 10.2196/30431. PMID 34435960